CLINICAL TRIAL: NCT01032148
Title: Phase I Study of LBH589, A Novel Oral Deacetylase Inhibitor in Patients With Recurrent or Refractory Hodgkin or Non-Hodgkin's Lymphoma
Brief Title: Study of LBH589, A Deacetylase Inhibitor in Patients With Recurrent or Refractory Hodgkin or Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPCI I 147408
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma
Keywords: Recurrent; Refractory
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Recurrence | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LBH589 (Experimental): LBH589 administered orally as once daily dose of 20 mg po q M, W, F on a q 28 day cycle, escalating to a maximum dase of 60 mg
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589 — LBH589 will be administered orally as once daily dose of 20 mg po q M, W, F on a q28 day cycle.

SUMMARY:
The purpose of this study is to find out the effects of a drug called LBH589 when given to people with recurrent or refractory Hodgkin or Non-Hodgkin's lymphoma. The safety of this drug will also be studied. The participants' physical state, changes in the size of the tumor, or state of Hodgkin or non-Hodgkin's Lymphoma, and laboratory findings taken while on-study will help the researchers decide if LBH589 is safe and effective.

DETAILED DESCRIPTION:
This is an open-label, standard 3-3 dose finding scheme with a modification that allows intra-patient dose modification to determine maximum tolerated dose and toxicity profile of LBH589 in patients with recurrent or refractory Hodgkin's or non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age ≥ 18 years old with relapsed/refractory Hodgkin lymphoma or NHL patients who have relapsed or are refractory after receiving a minimum of two prior therapies
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed

Laboratory requirements:

* ANC ≥ 1.5 x 10(9th)/L, unless due to bone marrow involvement with lymphoma
* Hemoglobin ≥ 9 g/dl without packed red blood cell dependency, unless due to bone marrow involvement with lymphoma
* Platelets ≥ 100 x 10(9th)/L, unless due to bone marrow involvement with lymphoma
* Serum creatinine ≤ 1.5 x Upper limit of Normal, or calculated Creatinine Clearance ≥ 50 mL/min
* AST and ALT ≤ 2.5 x Upper limit of Normal, unless due to liver involvement with lymphoma
* Serum bilirubin ≤ 1.5 x Upper limit of Normal
* Albumin > 3.0 g/dl
* Serum potassium ≥ Lower limit of Normal
* Total serum calcium [corrected for serum albumin] or ionized calcium ≥ Lower limits of normal
* Serum magnesium ≥ Lower limit of Normal
* Serum phosphorus ≥ Lower limit of Normal
* TSH ≥ LLN and free T4 within normal limits. Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
* Baseline MUGA or ECHO must demonstrate LVEF ≥ 50%
* ECOG Performance Status of ≤ 2

Exclusion Criteria:

* Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
* Patients who will need valproic acid for any medication during the study or within 5 days prior to first LBH589 treatment
* Peripheral neuropathy ≥ CTCAE grade 1
* Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:
* Patients with congenital QT syndrome
* History or presence of sustained ventricular tachyarrhythmia.
* Any history of ventricular fibrillation or torsade de pointes
* Bradycardia defined as Heart Rate < 50 bpm. Patients with pacemakers are eligible if Heart Rate ≥ 50 bpm
* Screening EKG with a QTc.450msec
* Right Bundle branch block + left anterior hemiblock (bifascicular block)
* Patients with myocardial infarction or unstable angina ≤ 6 months prior to starting study drug
* other clinically significant heart disease (e.g. CHF NY Heart Association class III or IV, uncontrolled hypertension, history of labile hypertension or history of poor compliance with an antihypertensive regimen)
* Impairment of GI function or GI disease that may significantly alter the absorption of LBH589
* Patients with Diarrhea > CTCAE grade 1
* Other concurrent severe and/or uncontrolled medical conditions (e.g. uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values that could cause unaccepted safety risks or compromise compliance with the protocol
* Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Concomitant use of CYP3A4 inhibitors
* Patients who have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites(which ever is longer) and who have not recovered from side effects of those therapies
* Patients who have received either immunotherapy within ≤ 8 weeks;chemotherapy within ≤ 4 weeks or radiation therapy to >30% of marrow-bearing bone within ≤ weeks prior to starting study treatment or who have not yet recovered from side effects of such therapies
* Patients with an active bleeding tendency or is receiving any treatment with therapeutic doses of sodium warfarin or coumadin derivatives. Low doses of Coumadin (e.g.≤2 mg/day) to maintain line patency is allowed.
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Women who are pregnant or breast feeding or women of childbearing potential not using effective method of birth control
* Male patients whose sexual partners are women of childbearing potential not using effective birth control
* Patients with prior malignancy within 5 years (except for basal or squamous cell carcinoma, in situ cancer of the cervix or early stage prostate or bladder carcinomas)
* Patients with known positivity for HIV or hepatitis C: baseline testing for HIV and Hepatitis C is not required
* Prior allogenic stem cell transplant
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff
* Patients taking CYP2D6 inhibitors should be carefully monitored, but these drugs are not necessarily contraindicated when use concomitantly with LBH. Use of these drugs is not an exclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose (MTD) of LBH589 | 2 years

SECONDARY OUTCOMES:
Determine toxicity profile in study population | 28 days after Cycle 2 Day 1
Determine anti-lymphoma activity of LBH589 in (non-CTCL) Hodgkin's and non-Hodgkin's lymphoma patients | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Hernandez, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States